CLINICAL TRIAL: NCT04788550
Title: A Prospective, Open Label, Randomized Control Trial to Study the Effect of Different Remineralizing Agents on White Spot Lesions and Dental Plaque During Orthodontic Retention
Brief Title: The Effect of Different Remineralizing Agents on White Spot Lesions and Dental Plaque During Orthodontic Retention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, Department of Paediatric Dentistry and Orthodontics, Faculty of Dentistry, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGD_190005
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Orthodontic Appliance Complication
Keywords: White Spot Lesion; Bacterial count( Streptococcus & Lactobacillus count); Salivary profile(salivary flow rate, buffering capacity, pH)
MeSH Terms: interventions — Sodium Fluoride; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: Group 1 The participants in group one will act as control group as they will be advised in using fluoridated toothpaste to brush twice daily during the follow up periods
  Group 2 The participants in this group will received fluoride varnish (5% sodium fluoride) treatment
  Group 3 The participants will be advised to use pea size CPP-ACP plus crème (900ppm fluoride)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toothpaste group (Active Comparator): Control group using fluoridated toothpaste
  Interventions: Combination Product: Fluoridated toothpaste
- Fluoride Varnish group (Experimental): Fluoride varnish (5% sodium fluoride) application on 3 months interval
  Interventions: Combination Product: fluoride varnish (5% sodium fluoride)
- CPP-ACP plus crème group (Experimental): CPP-ACP plus crème application 2 times daily
  Interventions: Combination Product: CPP-ACP plus crème group

INTERVENTIONS:
Combination Product: Fluoridated toothpaste — Group 1 will act as control group. Participants will be advised to brush twice daily using fluoridated toothpaste during the follow up periods. No other fluorides supplements will be allowed to use.
  Other Names: Colgate® Maximum cavity protection great regular flavour
  Arms: Toothpaste group
Combination Product: fluoride varnish (5% sodium fluoride) — Approximately 0.5-1.0ml fluoride varnish will be applied on the tooth surface (labially) with the paint-on method fom canines to canines. No other fluorides supplements will be allowed to use.
  Other Names: Colgate Duraphat 22,600 ppmF; 22,600 ppm Sodium Fluoride varnish
  Arms: Fluoride Varnish group
Combination Product: CPP-ACP plus crème group — Pea size CPP-ACP plus crème on the tooth surfaces using a clean fingers twice daily after brushing their teeth with fluoridated toothpaste. No other fluorides supplements will be allowed to use.
  Other Names: GC Tooth Mousse Plus®
  Arms: CPP-ACP plus crème group

SUMMARY:
Dental caries is a decay process that breaks down the tooth. The earliest clinical signs of active dental caries is seen as 'white spot lesions' (WSLs). WSLs causes porosity below the tooth surface as a result of demineralization that gives the lesion a milky white appearance.

Many WSLs persevere even a decade after orthodontic appliance removal and remain a cosmetic problem. After removal of fixed appliances, a considerable improvement of WSLs can be seen during the first 6-24 months, but the degree of improvement varies between individuals.

Two common bacteria in dental plaque causes caries: Streptococcus mutans (SM) and Lactobacillus acidophilus (LA) in the plaque contributes to the initiation and progression of caries, respectively.

A major strategy suggested to deal with existing WSL after debond is to facilitate remineralisation using remineralising agents that contain fluoride. This can be from daily use of fluoridated toothpastes or having additional dose of fluoride application. Certain agents also contain casein phosphopeptide-stabilize amorphous calcium phosphate (CPP-ACP) that is believed to have an antibacterial and buffering effect on plaque and interfere the growth and adherence of bacteria.

DETAILED DESCRIPTION:
Rationale of the study :

Currently there is insufficient evidence on the most effective regime of fluoride application to regress post orthodontic WSLs and how it affects the quality and quantity of oral microbial flora.

The study aims to determine the effect of different remineralizing agents on white spot lesions and dental plaque of post-orthodontic treatment patients.

The objectives are:

1. To compare the tooth surface changes (based on ICDAS, optical changes and patient perception) of white spot lesion treated with different remineralizing agents during orthodontic retention
2. To compare the bacterial count (including streptococcus and lactobacillus) in subjects with white spot lesions treated with different remineralizing agents during orthodontic retention
3. To compare the salivary profile (flow rate, Ph, buffering capacity) in subjects with white spot lesion treated with different remineralizing agents during orthodontic retention

Sample size calculation :

Sample size was calculated using G-power. Given an effect size of 0.49 (Jung et al., 2014), 80% power of study, alpha of 5% and 7 measurements, the sample size required was 27. With a 10% dropout, the final sample size is 30.

Methodology :

A. Subjects screening and preparation

Orthodontic patients treated with at least fixed appliances on the maxillary arch at the Faculty of Dentistry, University of Malaya whom are scheduled for debond, are invited to participate in this study. Participants will be screened for white spot lesions based on the inclusion and exclusion criteria. Participants will be randomly allocated to 3 groups that will receive remineralizing applications according to their allocated groups:

Group 1 The participants in group 1 will act as control group as they will be advised in using fluoridated toothpaste to brush twice daily during the follow up periods. No other fluorides supplements will be allowed to use.

Group 2 The participants in this group will received fluoride varnish (5% sodium fluoride) treatment. The labial surface of each tooth will be polished with non-fluoridated pumice powder and will be rinsed and dried thoroughly. Approximately 0.5-1.0ml fluoride varnish will be applied on the tooth surface (labially) with the paint-on method from canines to canines. After varnish application, patients will be advised not to drink for at least 30 minutes and not to brush teeth or eat food for the next 4 hours after application. Participants can brush teeth the night after application. The participants will be advised to brush their teeth daily with fluoridated toothpaste. Fluoride varnish application will be on 3 months intervals from first review visit (T1). No other fluorides supplements will be allowed to use.

Group 3 The participants will be advised to use pea size CPP-ACP plus crème on the tooth surfaces using a clean fingers twice daily following brushing their teeth with fluoridated toothpaste. The participants will be taught to keep the CPP-ACP plus crème on the tooth surface for at least 3 minutes before rinsing the mouth. After application of CPP-ACP plus crème, participants will be advised not to drink or eat for at least 30 minutes. No other fluoride supplements will be allowed to use.

During the first appointment (T0),

1. Debond procedure will be done according to the standard protocol.
2. Two sets of impression will be taken for the construction of study model, construction of the standard retainers and also for the research purpose.
3. Participants will be screen for white spot lesion by using the Optical Coherence Tomography (Santec) . A jig will be constructed for reproducible positioning of the probe. Two maxillary teeth with the worst WSL will be selected for each patient to measure the lesion depth and integrated refractivity. The intraoral photos of the maxillary teeth will be taken.
4. The salivary profile (flow rate, Ph, buffering capacity) will be measured using Saliva- Check BUFFER (GC America) according to the manufacturer's instruction.
5. Plaque samples will be collected with sterile swabs from the enamel surface of each tooth with the identified WSL to measure the bacterial count.

1 day after T0,

1. Participants will receive pressure formed or thermoplastic retainer in upper arch and instructed to wear their retainers all day (for at least 8 hours) and wear them after toothbrushing.
2. ICDAS score and optical changes (lesion depth and integrated refractivity) of the white spot lesion will be measured.
3. Participants will be given a set of questionnaires to assess the compliance to the remineralizing agent application and perception on the WSL.

Treatment follow up

1. The participants will be coordinated for follow up after 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), and 18 months (T5)
2. During the follow up visit , each participant will be subjected to the measurement of :

   * tooth surface changes
   * bacterial count
   * salivary profile
   * intraoral photos of maxillary teeth
3. Participants will be given a set of questionnaires at every follow up visit to assess the compliance to the application of remineralizing agent and perception of the WSLs

Statistical Analysis

Data analysis will be done using the SPSS version 22. Descriptive date will be expressed as mean ± standard deviation (SD) unless otherwise stated. Repeated measurement ANOVA will be used for analysis of normally distributed variables. Kruskal-Wallis ANOVA will be used for non-normally distributed data. A value of P < 0.05 is considered statistically significant. The data collected will be analyzed using an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on multibracket fixed appliance treatment
* Subjects with 2 or more bracketed surfaces with labial subsurface WSLs from
* upper right permanent canine (13) to upper left permanent canine (23) with an ICDAS II score of 1 and 2 will be selected.
* Indicated for thermoform or vacuum formed retainers on the upper arch.

Exclusion Criteria:

* Systemic diseases or any physical anomalies.
* Subjects with intention to move out from Klang Valley area for the next 1.5 years.
* Periodontal diseases (pocket depth of more than 3mm).
* Smoker.
* Severe fluorosis or any enamel abnormalities.
* Antimicrobial agents or antibiotic therapy within the past 3 months.
* Orthognathic surgery cases, cleft lip and palate.
* Single arched lower fixed orthodontic treatment.
* Milk protein and benzoate preservatives (a common preservatives) allergies.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ICDAS score of the white spot lesion. | 18 months
  Changes in WSL measured based on ICDAS score :
  * 0 No evidence of caries
  * 1 Initial caries
  * 2 Distinct visual change in enamel
  * 3 Localised enamel breakdown due to caries with no visible dentine
  * 4 Underlying dark shadow from dentine
  * 5 Distinct cavity with visible dentine
  * 6 Extensive distinct cavity with visible dentine
Optical changes (refractive index) of the white spot lesion. | 18 months
  Changes in WSL measured in lesion depths (LD in μm).
Patient perception of the WSL | 18 months
  Patient will be given a set of questionnaires at every follow up visit to assess the
  1. Compliance to the remineralizing agent application
  2. Perception on the WSL
  The perception will be based on the Likert scale
Dental plaque total bacterial count, Streptococcus count, Lactobacillus count. | 18 months
  Plaque samples will be collected with sterile swabs from the enamel surface of each tooth with the identified WSL to measure the bacterial count.
  The colony forming units of each plates is enumerated and the cfu/mL will be calculated

SECONDARY OUTCOMES:
Salivary profile (salivary flow rate) | 18 months
  The stimulated saliva will be collected by having the subject spit for 10 minutes into a sterile plastic graduated cup with 1-mL gradation marks Collected salivary volume was measured in millilitres, and salivary flow rate was calculated based on a collection time of 10 minutes (millilitres per minute).
Salivary profile (buffering capacity) | 18 months
  The saliva buffer capacity will be measured using strips (Saliva-Check BUFFER) and measured against standards assigned by the manufacturer Using a pipette, a saliva sample will be taken, and 1 drop will be placed on each of the 3 test pads. Test pads will change colour immediately, but the final colour will only detect after 2 minutes.
  Then the result will be calculated by adding the points according to the final colour of each pad.
  * green - 4 points
  * green/ blue - 3 points
  * blue - 2 points
  * red/blue - 1 point
  * red - 0 points
  All points were counted, and result was determined:
  * 0 - 5 points as very low buffering ability,
  * 6 - 9 points as low,
  * 10 - 12 points as normal/high.
  The buffering capacity is based on total points , 0-5 ( very low) , 6-9 (low), 10-12 (normal)
Salivary profile (pH) | 18 months
  The pH test strip will be placed inside the saliva collection cup for 10 seconds.
  The colour of the strip will be compared to the testing chart available in the kit .

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Orthodontic Clinic, Faculty Of Dentistry, University Of Malaya, Kuala Lumpur, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pitts NB, Zero DT, Marsh PD, Ekstrand K, Weintraub JA, Ramos-Gomez F, Tagami J, Twetman S, Tsakos G, Ismail A. Dental caries. Nat Rev Dis Primers. 2017 May 25;3:17030. doi: 10.1038/nrdp.2017.30. PMID 28540937
- [Background] Simon-Soro A, Mira A. Solving the etiology of dental caries. Trends Microbiol. 2015 Feb;23(2):76-82. doi: 10.1016/j.tim.2014.10.010. Epub 2014 Nov 27. PMID 25435135
- [Background] van Houte J. Role of micro-organisms in caries etiology. J Dent Res. 1994 Mar;73(3):672-81. doi: 10.1177/00220345940730031301. PMID 8163737
- [Background] Mizrahi E. Enamel demineralization following orthodontic treatment. Am J Orthod. 1982 Jul;82(1):62-7. doi: 10.1016/0002-9416(82)90548-6. PMID 6984291
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Ogaard B, Rolla G, Arends J, ten Cate JM. Orthodontic appliances and enamel demineralization. Part 2. Prevention and treatment of lesions. Am J Orthod Dentofacial Orthop. 1988 Aug;94(2):123-8. doi: 10.1016/0889-5406(88)90360-5. PMID 3165239
- [Background] Mitchell L. Decalcification during orthodontic treatment with fixed appliances--an overview. Br J Orthod. 1992 Aug;19(3):199-205. doi: 10.1179/bjo.19.3.199. No abstract available. PMID 1390575
- [Background] Artun J, Brobakken BO. Prevalence of carious white spots after orthodontic treatment with multibonded appliances. Eur J Orthod. 1986 Nov;8(4):229-34. doi: 10.1093/ejo/8.4.229. No abstract available. PMID 3466795
- [Background] Gwinnett AJ, Ceen RF. Plaque distribution on bonded brackets: a scanning microscope study. Am J Orthod. 1979 Jun;75(6):667-77. doi: 10.1016/0002-9416(79)90098-8. No abstract available. PMID 377979
- [Background] Chapman JA, Roberts WE, Eckert GJ, Kula KS, Gonzalez-Cabezas C. Risk factors for incidence and severity of white spot lesions during treatment with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):188-94. doi: 10.1016/j.ajodo.2008.10.019. PMID 20691360
- [Background] Featherstone JD. The science and practice of caries prevention. J Am Dent Assoc. 2000 Jul;131(7):887-99. doi: 10.14219/jada.archive.2000.0307. PMID 10916327
- [Background] Chatterjee R, Kleinberg I. Effect of orthodontic band placement on the chemical composition of human incisor tooth plaque. Arch Oral Biol. 1979;24(2):97-100. doi: 10.1016/0003-9969(79)90056-6. No abstract available. PMID 45361
- [Background] Scheie AA, Arneberg P, Krogstad O. Effect of orthodontic treatment on prevalence of Streptococcus mutans in plaque and saliva. Scand J Dent Res. 1984 Jun;92(3):211-7. doi: 10.1111/j.1600-0722.1984.tb00881.x. PMID 6589736
- [Background] Freitas AO, Marquezan M, Nojima Mda C, Alviano DS, Maia LC. The influence of orthodontic fixed appliances on the oral microbiota: a systematic review. Dental Press J Orthod. 2014 Mar-Apr;19(2):46-55. doi: 10.1590/2176-9451.19.2.046-055.oar. PMID 24945514
- [Background] Nyvad B. Microbial colonization of human tooth surfaces. APMIS Suppl. 1993;32:1-45. No abstract available. PMID 8494649
- [Background] Socransky SS, Manganiello SD. The oral microbiota of man from birth to senility. J Periodontol. 1971 Aug;42(8):485-96. doi: 10.1902/jop.1971.42.8.485. No abstract available. PMID 4998039
- [Background] Lara-Carrillo E, Montiel-Bastida NM, Sanchez-Perez L, Alanis-Tavira J. Effect of orthodontic treatment on saliva, plaque and the levels of Streptococcus mutans and Lactobacillus. Med Oral Patol Oral Cir Bucal. 2010 Nov 1;15(6):e924-9. doi: 10.4317/medoral.15.e924. PMID 20383105
- [Background] Schirrmeister JF, Gebrande JP, Altenburger MJ, Monting JS, Hellwig E. Effect of dentifrice containing 5000 ppm fluoride on non-cavitated fissure carious lesions in vivo after 2 weeks. Am J Dent. 2007 Aug;20(4):212-6. PMID 17907481
- [Background] Alexander SA, Ripa LW. Effects of self-applied topical fluoride preparations in orthodontic patients. Angle Orthod. 2000 Dec;70(6):424-30. doi: 10.1043/0003-3219(2000)0702.0.CO;2. PMID 11138645
- [Background] Shungin D, Olsson AI, Persson M. Orthodontic treatment-related white spot lesions: a 14-year prospective quantitative follow-up, including bonding material assessment. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):136.e1-8; discussion 136-7. doi: 10.1016/j.ajodo.2009.05.020. PMID 20691346
- [Background] Rosenbloom RG, Tinanoff N. Salivary Streptococcus mutans levels in patients before, during, and after orthodontic treatment. Am J Orthod Dentofacial Orthop. 1991 Jul;100(1):35-7. doi: 10.1016/0889-5406(91)70046-Y. PMID 2069145
- [Background] Duggal MS, van Loveren C. Dental considerations for dietary counselling. Int Dent J. 2001;51(6 Suppl 1):408-12. doi: 10.1111/j.1875-595x.2001.tb00588.x. PMID 11794563
- [Background] Marshall TA. Chairside diet assessment of caries risk. J Am Dent Assoc. 2009 Jun;140(6):670-4. doi: 10.14219/jada.archive.2009.0252. PMID 19491162
- [Background] Ogaard B. Effects of fluoride on caries development and progression in vivo. J Dent Res. 1990 Feb;69 Spec No:813-9; discussion 820-3. doi: 10.1177/00220345900690S155. PMID 2179345
- [Background] Knosel M, Attin R, Becker K, Attin T. External bleaching effect on the color and luminosity of inactive white-spot lesions after fixed orthodontic appliances. Angle Orthod. 2007 Jul;77(4):646-52. doi: 10.2319/060106-224. PMID 17605483
- [Background] Baysan A, Lynch E, Ellwood R, Davies R, Petersson L, Borsboom P. Reversal of primary root caries using dentifrices containing 5,000 and 1,100 ppm fluoride. Caries Res. 2001 Jan-Feb;35(1):41-6. doi: 10.1159/000047429. PMID 11125195
- [Background] Reynolds EC. The prevention of sub-surface demineralization of bovine enamel and change in plaque composition by casein in an intra-oral model. J Dent Res. 1987 Jun;66(6):1120-7. doi: 10.1177/00220345870660060601. PMID 3476583
- [Background] Selwitz RH, Ismail AI, Pitts NB. Dental caries. Lancet. 2007 Jan 6;369(9555):51-9. doi: 10.1016/S0140-6736(07)60031-2. PMID 17208642
- [Background] Sitthisettapong T, Doi T, Nishida Y, Kambara M, Phantumvanit P. Effect of CPP-ACP Paste on Enamel Carious Lesion of Primary Upper Anterior Teeth Assessed by Quantitative Light-Induced Fluorescence: A One-Year Clinical Trial. Caries Res. 2015;49(4):434-41. doi: 10.1159/000434728. Epub 2015 Jul 29. PMID 26228178
- [Background] Davidson CL, Bekke-Hoekstra IS. The resistance of superficially sealed enamel to wear and carious attack in vitro. J Oral Rehabil. 1980 Jul;7(4):299-305. doi: 10.1111/j.1365-2842.1980.tb00448.x. PMID 6931880
- [Background] Hochli D, Hersberger-Zurfluh M, Papageorgiou SN, Eliades T. Interventions for orthodontically induced white spot lesions: a systematic review and meta-analysis. Eur J Orthod. 2017 Apr 1;39(2):122-133. doi: 10.1093/ejo/cjw065. PMID 27907894
- [Derived] Wan Hassan WN, Tee YY, Md Razali K, Abdul Razak AA, Lim HH, Zakaria N, Sukumaran P, Mohd Tahir NNZ, Chew HP. A 12-months randomized clinical trial comparing fluoride-based remineralising protocols on post-orthodontic initial caries lesions. Clin Oral Investig. 2025 Feb 5;29(2):111. doi: 10.1007/s00784-025-06172-0. PMID 39907699